CLINICAL TRIAL: NCT02398136
Title: Randomized Controlled Trial of Repeated Dose Ketamine in Post Traumatic Stress Disorder (PTSD)
Brief Title: To Test the Potential Efficacy of Repeated Intranasal Administration of Ketamine as a Treatment for PTSD
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: FDA and IRB recommended different mode of medication administration
Sponsor: Adriana Feder (Other)
Responsible Party: Sponsor-Investigator, Adriana Feder, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 14-1781
Record Dates: First submitted 2014-11-07; First posted 2015-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: PTSD
Keywords: intervention; ketamine; PTSD; treatment; posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Intranasal ketamine up to 75 mg, delivered over 20 minutes, frequency: 3x/week for 4 weeks.
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): Intranasal midazolam 3.75mg, delivered over 20 minutes, frequency: 3x/week for 4 weeks.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine
  Other Names: Intranasal ketamine
  Arms: Ketamine
Drug: Midazolam
  Other Names: Placebo
  Arms: Midazolam

SUMMARY:
The purpose of this study is to see whether ketamine, when given repeatedly via the nose (intranasally), can produce a quick and persistent improvement in PTSD symptoms. At higher doses, ketamine has been used for many years as an anesthetic for medical procedures, and at lower doses may be an effective treatment in patients with major depression and PTSD.

DETAILED DESCRIPTION:
The objective of the present research protocol, a parallel-arm, double-blind, randomized controlled clinical trial, is to test the efficacy of repeated intranasal administration of the glutamatergic NMDA receptor antagonist ketamine in providing (1) rapid relief of and (2) sustained improvement in core PTSD symptoms and co-morbid depressive symptoms in patients with chronic PTSD. The effects of ketamine will be compared with those of repeated intranasal administration of the benzodiazepine anesthetic midazolam, which mimics some of the acute subjective effects of ketamine but is expected to have lesser or less sustained anxiolytic effect, and no sustained antidepressant effect.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18-65 years of age;
* Participants must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign a written informed consent document;
* Participants must fulfill DSM-5 criteria for current civilian or combat-related PTSD, based on clinical assessment by a study psychiatrist and on the CAPS -this is done to ensure at least moderate severity and to safeguard against high placebo response rates;
* Women must be using a medically accepted reliable means of contraception (if using an oral contraceptive medication, they must also be using a barrier contraceptive) or not be of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year);
* Women of childbearing potential must have a negative pregnancy test at screening and prior to each intranasal administration;
* Participants must be able to identify a family member, physician, or friend (i.e. someone who knows them well) who will participate in a Treatment Contract (and e.g. contact the study physician on their behalf in case manic symptoms or suicidal thoughts develop).

Exclusion Criteria:

* Women who plan to become pregnant, are pregnant or are breast-feeding (because the medical risk of using ketamine during pregnancy and breast-feeding is unknown);
* Serious, unstable medical illnesses such as hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease, including gastro-esophageal reflux disease, obstructive sleep apnea, history of difficulty with airway management during previous anesthetics, ischemic heart disease and uncontrolled hypertension, and history of severe head injury;
* Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG;
* Patients with uncorrected hypothyroidism or hyperthyroidism;
* Hormonal treatment (e.g., estrogen) started in the 3 months prior to the first intranasal administration day;
* Use of evidence-based individual psychotherapy (such as prolonged exposure) during the study;
* History of autism, mental retardation, pervasive developmental disorders, or Tourette's syndrome;
* History of one or more seizures without a clear and resolved etiology;
* History of (hypo)mania;
* Past or current presence of psychotic symptoms, or diagnosis of a lifetime psychotic disorder including schizophrenia or schizoaffective disorder;
* Drug or alcohol abuse or dependence within the preceding 3 months; a rather narrow time period was chosen, however, in order to allow participation by individuals with a history of substance abuse or dependence problems that could be secondary to their PTSD, and to more closely approximate patients seen in real-world settings; this is the same period of time that we used in our recently completed study of IV ketamine for PTSD.
* Previous recreational use of ketamine or PCP;
* Current diagnosis of bulimia nervosa or anorexia nervosa;
* Diagnosis of schizotypal or antisocial personality disorder (since these are known to reduce the possibility of study completion); other Axis II diagnoses will be allowed;
* Patients judged clinically to be at serious and imminent suicidal or homicidal risk.
* A blood pressure of one reading over 160/90 or two separate readings over 140/90 at screen or baseline visits
* Patients who report current treatment with a benzodiazepine, an opioid medication, or a mood stabilizer (such as valproic acid or lithium) within 2 weeks prior to randomization; patients taking stable doses of antidepressant medication for 3 months prior to randomization will be allowed.
* For subjects who may participate in the MRI portion of the study, claustrophobia, any trauma or surgery which may have left magnetic material in the body, magnetic implants or pacemakers, and inability to lie still for 1 hour or more.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Impact of Events Scale-Revised (IES-R) | 24 hours
  The IES-R is used to self-report measures of stress reactions to traumatic events. It measures both intrusion and avoidance.

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | up to 4 weeks
  The CAPS is a structured clinical interview designed to assess the essential features of PTSD.
Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR) | 24 hours
  The QIDS-SR is a 16-item self-rated instrument designed to assess the severity of depressive symptoms present in the past seven days.
Montgomery Asberg Depression Rating Scale (MADRS) | 24 hours
  The MADRS is a 10-item instrument used for the evaluation of depressive symptoms and for the assessment of any changes to those symptoms.
Patient-Rated Inventory of Side Effects (PRISE) | 24 hours
  PRISE is a 7-item self report used to qualify side effects by identifying and evaluating the tolerability of each symptoms.
Sheehan Disability Scale (SDS) | 24 hours
  The SDS is a 10 point visual analog scale developed to assess functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Feder, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai